CLINICAL TRIAL: NCT07178470
Title: Concordance and Discordance in the Assessment of Volume Status in Home Dialysis Patients: A Comparison of Modified Medical Research Council Dyspnea Scale, Physical Exam, and Point of Care Ultrasound (POCUS)
Status: Not yet recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nupur Gupta, Associate Professor of Clinical Medicine, Indiana University
Other Study IDs: 28387
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Fluid Overload; POCUS; Lung Ultrasound; Volume Status
Keywords: pocus; fluid overload; lung ultrasound; volume status; modified Medical Research Council Dyspnea Scale; mMRC dyspnea scale
MeSH Terms: conditions — Edema | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Only a single cohort/group: This study includes only one group all of whom get the same testing
  Interventions: Diagnostic Test: Modified Medical Research Council (mMRC) Dyspnea scale , , point-of-care ultrasound (POCUS), specifically lung ultrasound (LUS) and physical examination

INTERVENTIONS:
Diagnostic Test: Modified Medical Research Council (mMRC) Dyspnea scale , , point-of-care ultrasound (POCUS), specifically lung ultrasound (LUS) and physical examination — After obtaining informed consent, the Modified Medical Research Council (mMRC) Dyspnea scale will be administered to patients, and their responses will be recorded on a scale of 0 to +4. During the same clinical visit, a physical examination will be performed by the primary nephrologist, who will categorize the patient's volume status as hypovolemic, euvolemic, mild, moderate, or severe volume overloaded. Finally, point-of-care ultrasound (POCUS), specifically lung ultrasound (LUS), will be performed. Patients will be assigned a score based on the number of B-lines observed. We will measure discordance and concordance between the LUS and physical exam, the LUS and mMRC dyspnea scale, and between the physical exam and mMRc dyspnea scale.
  Other Names: Ultrasound device either Phillips or Butterfly

SUMMARY:
Fluid overload, which is when your body has too much fluid, is one of the reasons why people on home dialysis need to go to the hospital. Fluid overload (when body has too much fluid) commonly presents as trouble breathing and leg swelling. Traditionally, doctors check for this by asking patients if they have any symptoms like leg swelling or shortness of breath and by doing a physical exam which includes listening to the lungs or looking for swelling in legs. However, a newer, safe, and non-invasive method called point-of-care ultrasound (POCUS) has become very popular. However, we don't have a lot of research yet on how POCUS and LUS (lung ultrasound) specifically help home dialysis patients, including those on peritoneal dialysis or home hemodialysis. Peritoneal dialysis is a way to clean your blood by putting a special fluid into your belly through a small tube. The fluid uses the natural lining of your belly as a filter to remove waste and extra water. Home hemodialysis is a treatment where a machine acts like an artificial kidney to clean your blood. You get trained to do this yourself at home by connecting to the machine with a couple of needles, which cleans your blood of waste and extra fluid. POCUS, especially a (LUS), has been shown to be useful for dialysis patients in outpatient units.

This study will compare different 3 different methods of detecting fluid overload: answering various survey questions, completing a physical exam, and a LUS. The study seeks to determine which of these methods is the best method to determine fluid overload.

You were selected as a possible participant because you are over 18 years old, diagnosed with End-stage kidney disease, and have been receiving home dialysis for at least three months.

DETAILED DESCRIPTION:
This study involves collecting information about you or from you. If you agree to be in the study, you will do your best to complete the following:

* Provide consent for us to review your medical records, including those from your dialysis center.
* The entire study visit will last for approximately 30-60 minutes including checking blood pressure, weight, questionnaire, doctor's visit and ultrasound
* We will measure blood pressure and weight if it's a part of your routine visit
* You will be given a questionnaire called modified medical research council dyspnea scale which includes only 1 question and anticipated to take less than a minute to answer
* After this, you will have your visit with your kidney doctor as usual. The doctor will assess how much excess fluid you might have by listening to your lungs and checking for swelling in your legs. They will not be given the results of the above survey.

After this, you'll go to a private room for the ultrasound procedure:

You'll lie flat on your back, and we'll expose your chest. A small amount of gel will be put on your skin, and we'll use a handheld ultrasound device to lightly press on your chest. We'll scan eight specific areas on your chest (four on each side) to look for something called "B-lines," which can show if there's extra fluid in your lungs. This ultrasound part of the visit should only take about 10 to 15 minutes in total.

Care will be taken to expose only the area being scanned. A chaperone (someone else in the room) will be present for all female patients. All male patients will be asked if they want a chaperone. If they say yes, a chaperone will be present during the ultrasound procedure. After the ultrasound, we'll wipe off the gel with a cloth, and you'll be ready to leave the room.

We expect the entire study from enrollment to the completion of data collection for all subjects, to last 9 months. However, your study visit will last only for 30-60minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Greater than 18 years.
2. Diagnosis: End-stage kidney disease (ESKD).
3. Treatment: Receiving home dialysis, either peritoneal dialysis (PD) or home hemodialysis (HHD).
4. Duration of Home Dialysis: At least three months on home dialysis.

Exclusion Criteria:

1. Consent: Inability to provide informed consent.
2. Inclusion Criteria: Not meeting any of the inclusion criteria.
3. Pregnancy.
4. Urgent-Start PD.
5. Any other obvious cause of shortness of breath not related to volume overload including but not limited to pneumonia, pneumothorax, advanced COPD and Interstitial lung disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All home dialysis patient's at DaVita Home Dialysis of Indianapolis who are on home dialysis including peritoneal and home hemodialysis will be potential candidates
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Discordance and concordance between the LUS and physical exam, the LUS and mMRC dyspnea scale, and between the physical exam and mMRc dyspnea scale. | 6-12 months
  We will measure discordance and concordance between the LUS and physical exam, the LUS and mMRC dyspnea scale, and between the physical exam and mMRc dyspnea scale. A pair is concordant if the observation ranking higher on one variable also ranks higher on the second measure. The pair is discordant if the observation ranking higher on one endpoint measure and ranks lower on the other. The pair is tied if the subjects have the same classification on both measures. Depending on the results additional analyses may be conducted to determine differences between peritoneal dialysis and home hemodialysis, or differences by sex, or differences by those on or off diuretics on those with and without residual renal function assessed by 24 hour urine output routinely done as part of standard care for the PD patients
discordance and concordance between the LUS and physical exam, the LUS and mMRC dyspnea scale, and between the physical exam and mMRc dyspnea scale. | Each participant will be involved in the study for 30-60 minutes which will include the questionnaire, physical examination, blood pressure, weight and ultrasound procedure.
  A pair is concordant if the observation ranking higher on one variable also ranks higher on the second measure. The pair is discordant if the observation ranking higher on one endpoint measure and ranks lower on the other. The pair is tied if the subjects have the same classification on both measures.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leidi A, Soret G, Mann T, Koegler F, Coen M, Leszek A, Dubouchet L, Guillermin A, Kaddour M, Rouyer F, Combescure C, Carballo S, Reny JL, Marti C, Stirnemann J, Grosgurin O. Eight versus 28-point lung ultrasonography in moderate acute heart failure: a prospective comparative study. Intern Emerg Med. 2022 Aug;17(5):1375-1383. doi: 10.1007/s11739-022-02943-9. Epub 2022 Feb 18. PMID 35181839
- [Background] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Background] Alexandrou ME, Theodorakopoulou MP, Sarafidis PA. Lung Ultrasound as a Tool to Evaluate Fluid Accumulation in Dialysis Patients. Kidney Blood Press Res. 2022;47(3):163-176. doi: 10.1159/000521691. Epub 2022 Jan 10. PMID 35008093
- [Background] Maw AM, Hassanin A, Ho PM, McInnes MDF, Moss A, Juarez-Colunga E, Soni NJ, Miglioranza MH, Platz E, DeSanto K, Sertich AP, Salame G, Daugherty SL. Diagnostic Accuracy of Point-of-Care Lung Ultrasonography and Chest Radiography in Adults With Symptoms Suggestive of Acute Decompensated Heart Failure: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Mar 1;2(3):e190703. doi: 10.1001/jamanetworkopen.2019.0703. PMID 30874784
- [Background] van Eck van der Sluijs A, Bonenkamp AA, van Wallene VA, Hoekstra T, Lissenberg-Witte BI, Dekker FW, van Ittersum FJ, Verhaar MC, van Jaarsveld BC, Abrahams AC; DOMESTICO study group. Differences in hospitalisation between peritoneal dialysis and haemodialysis patients. Eur J Clin Invest. 2022 Jun;52(6):e13758. doi: 10.1111/eci.13758. Epub 2022 Feb 15. PMID 35129213